CLINICAL TRIAL: NCT05751577
Title: TRanscatheter Aortic-Valve Implantation With or Without On-site Cardiac Surgery: the TRACS Trial
Acronym: TRACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government); Università degli Studi di Ferrara (Other); University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40-2023-SPER-AUSLBO
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Aortic Stenosis, Severe
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: TRACS is an all-comer, prospective, randomized, multicenter, open-label trial with blinded adjudicated evaluation of outcomes (PROBE)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL ARM: TAVI WITHOUT ON-SITE SURGERY (Experimental): After randomization, study TAVI operators of the participating center will schedule the patient for TAVI in their hospital without on-site surgery
  Interventions: Procedure: TAVI WITHOUT ON-SITE SURGERY
- CONTROL ARM: TAVI WITH ON-SITE SURGERY (Active Comparator): After randomization, the patient will immediately be placed on the waiting list of the referring center with on-site cardiac surgery. Study TAVI operators of the participating center will perform the TAVI procedure in the hospital with on-site surgery according to the waiting list schedule of the latter
  Interventions: Procedure: TAVI WITH ON-SITE SURGERY

INTERVENTIONS:
Procedure: TAVI WITHOUT ON-SITE SURGERY — After randomization, study TAVI operators of the participating center will schedule the patient for TAVI in their hospital without on-site surgery
  Arms: EXPERIMENTAL ARM: TAVI WITHOUT ON-SITE SURGERY
Procedure: TAVI WITH ON-SITE SURGERY — After randomization, the patient will immediately be placed on the waiting list of the referring center with on-site cardiac surgery. Study TAVI operators of the participating center will perform the TAVI procedure in the hospital with on-site surgery according to the waiting list schedule of the latter
  Arms: CONTROL ARM: TAVI WITH ON-SITE SURGERY

SUMMARY:
The primary efficacy objective is to determine whether a TAVI procedure performed by experienced operators in centers without on-site cardiac surgery is noninferior to TAVI procedure performed by the same operators in centers with on-site cardiac surgery in terms of all-cause death, stroke and rehospitalization for cardiovascular cause. The primary safety objective is to demonstrate that mortality associated with periprocedural complications actionable by emergent cardiac surgery did not differ between study arms.

DETAILED DESCRIPTION:
TRACS is an all-comer, prospective, randomized, multicenter, open-label trial with blinded adjudicated evaluation of outcomes (PROBE). The TRACS trial will involve centers without on-site cardiac surgery, but with experienced operators already performing TAVI at the referring center with on-site cardiac surgery. Thus, participating centers and their study TAVI operators must follow selective criteria for eligibility. Participants will be recruited after Heart Team indication to TAVI procedure. The eligibility of each single patient to the study MUST BE CONFIRMED and VALIDATED by unanimous decision of the Heart Team. Study patients will be randomized in a 2:1 fashion to TAVI procedure performed by the same experienced operators either in the center without on-site cardiac surgery or in the referring center with on-site cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis
* Indication to TAVI confirmed by the Study Heart Team

AND one of the following:

* Inoperable due to prohibitive operative risk
* High surgical risk as defined as STS score >8%

The presence of at least one clinical factor that, by unanimous judgment of the Study Heart Team, compromises the benefit/risk ratio in the case of emergent cardiac surgery:

* Porcelain aorta or severely atherosclerotic aorta
* Frailty/Reduced physical performance
* Cognitive impairment, dementia, or Parkinson's disease
* Severe liver disease/cirrhosis
* Hostile chest
* Internal mammalian artery or other critical conduit(s) crossing midline and/or adhering to the posterior table of the sternum
* Severe pulmonary hypertension and/or severe right ventricular dysfunction
* Severe Chronic Obstructive Pulmonary Disease (COPD)
* Age ≥85 years

Exclusion Criteria:

* Unsuitable for transfemoral TAVI
* Emergent TAVI
* Noncardiovascular comorbidity reducing life expectancy to <1 year
* Any factor precluding 1-year follow-up
* Refusal informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 1-year
  1-year cumulative occurrence of all-cause death, stroke and hospital readmission for CV cause To test if the outcome of TAVI procedures performed by experienced operators in the center without onsite cardiac surgery is non inferior to that of TAVI procedures performed by the same team in the center with on-site cardiac surgery
Primary safety endpoint | 1-year
  To test whether mortality due to periprocedural complications actionable by emergent cardiac surgery differs between the TAVI procedures performed in the center without on-site cardiac surgery and the TAVI procedures performed by the same team in the center with on-site cardiac surgery

SECONDARY OUTCOMES:
Secondary efficacy endpoints | 1-year
  All-cause death Cardiovascular death Myocardial infarction Hospital admission for cardiovascular cause Hospital admission for heart failure Cerebrovascular accident Ischemic stroke Hospital admission for pneumonia (± respiratory failure) Need for balloon aortic valvuloplasty for emergent condition Quality of life measured with the Eq-5D and KCCQ-12 scales Time spent on the waiting list before TAVI
Other safety endpoints | 1-year
  Cardiac tamponade Bleeding Kidney failure (requirement for renal replacement therapy) Severe aortic regurgitation (aortic regurgitation according to current guidelines) Multiorgan failure (failure of at least two organ systems) Vascular access site and access related complications Conduction disturbances and arrhythmias Endocarditis Valve thrombosis Valve malpositioning Valve embolization Ectopic valve deployment TAV-in-TAV deployment

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Ospedale San Donato di Arezzo, Arezzo
  - Ospedale Cardinal Massaia di Asti, Asti
  - Ospedale degli Infermi di Biella, Biella
  - Azienda Unità Sanitaria Locale, Bologna
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - Ospedale Misericordia di Grosseto, Grosseto
  - Azienda ULSS 3 Serenissima, Ospedale di Mirano, Mirano
  - Ospedale Guglielmo da Saliceto di Piacenza, Piacenza
  - Azienda Ospedaliera di Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannopollo G, Cocco M, Leone A, Sacca S, Mangino D, Picchi A, Reccia MR, Fineschi M, Meliga E, Audo A, Nobile G, Tumscitz C, Penzo C, Saia F, Rubboli A, Moretti C, Vignali L, Niccoli G, Cimaglia P, Rognoni A, Aschieri D, Iaccarino D, Ottani F, Cavazza C, Varbella F, Secco GG, Bolognese L, Limbruno U, Guiducci V, Campo G, Casella G. Transcatheter aortic-valve implantation with or without on-site cardiac surgery: The TRACS trial. Am Heart J. 2025 Feb;280:7-17. doi: 10.1016/j.ahj.2024.10.019. Epub 2024 Nov 4. PMID 39505122